CLINICAL TRIAL: NCT01416558
Title: A Multicenter Non-randomized Phase II Study to Evaluate Nab-paclitaxel in Metastatic Brest Cancer Patients Failing a Solvent Based Taxane as (Neo-)Adjuvant Treatment (Tiffany)
Brief Title: Nab-paclitaxel in Metastatic Breast Cancer Patients Failing Solvent Based Taxane (Tiffany)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated because of extrem low recruitment
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBG 65; 2011-000075-13 (EudraCT Number)
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Metastatic Breast Cancer
Keywords: German Breast Group; GBG Forschungs GmbH; GBG; GBG 65; Tiffany; Breast Cancer; Metastatic Breast Cancer; Nab-Paclitaxel; Abraxane; Taxane Failure
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nab-Paclitaxel — Nab-Paclitaxel 125 mg/m2 i.v. over 30 min. weekly in 5 out of 6 weeks
  Given until progression, unacceptable toxicity, patient's request or withdrawal from Study
  Other Names: Abraxane, EU/1/07/428/001

SUMMARY:
Nab-paclitaxel has demonstrated to be an active agent in breast cancer and probably a less toxic alternative to solvent based taxanes. It is indicated in metastatic breast cancer after failure of anthracyclines. However, most patients receive anthracyclines as well as taxanes as part of their (neo-)adjuvant therapy. There is currently no standard treatment for patients with an early relapse (<12 months) after a taxane containing (neo-)adjuvant therapy. Nab-paclitaxel, a novel nano-particle encapsulated paclitaxel is expected to have only limited cross-resistant to solvent-based taxanes and might therefore be indicated in this setting.

DETAILED DESCRIPTION:
Primary Objective:

To determine overall response rate (ORR) and to exclude that it is 20% or lower.

Secondary Objectives:

1. To determine compliance and toxicity of the therapy.
2. To determine clinical benefit rate (CBR) in patients with measurable disease.
3. To determine duration of response.
4. To determine progression-free survival (PFS).
5. To determine overall survival.
6. To assess biomarkers, e.g. SPARC expression in the tissue of the primary or metastatic tumor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
* Complete baseline documentation must be submitted via the web-based data collection system MedCODES to the GBG Forschungs GmbH.
* Diagnosis of locally advanced or metastatic hormone-sensitive or insensitive, HER2-negative or -positive breast cancer.
* Relapse within ≤ 12 months after completing (last day of last cycle) (neo-) adjuvant chemotherapy.
* Documented relapse of either a measurable or a non-measurable lesion according to the modified RECIST criteria.
* Previous neoadjuvant or adjuvant treatment with a solvent based taxane (paclitaxel or docetaxel) irrespective of dose and duration.
* Prior endocrine treatment for metastatic / advanced disease is allowed.
* Complete radiological and clinical tumor assessment within 4 weeks prior to registration performed as clinically indicated.
* Age ≥ 18 years.
* ECOG Performance Status ≤ 2 (irrespective of restrictions due to breast cancer).
* Laboratory requirements:Absolute neutrophil count (ANC) >= 1.5 x 109/L., Platelets >= 100 x 109/L., Hemoglobin >= 9 g/dL (>= 5.6 mmol/L)., Prothrombin time (PT) or international normalized ratio (INR) <= 1.2x ULN (upper normal limit), Partial thromboplastin time (PTT) <= 1.2x ULN, Total bilirubin < 1.5x ULN, ASAT (SGOT) and ALAT (SGPT) <= 2.5x ULN (concomitant elevations in serum bilirubin and ASAT/ALAT above 1.0x ULN are not permitted), Creatinine clearance >= 50 mL/min), Urine Protein to Creatinine Ratio (UPC) < 1 (if UPC >= 1, then 24-hour urine protein must be < 1 g).
* Normal cardiac function confirmed by ECG.
* A female either of: 1) Non-childbearing potential, i.e. physiologically incapable of becoming pregnant because of history of hysterectomy, bilateral oophorectomy (ovariectomy), bilateral tubal ligation or postmenopausal status.

  2) Childbearing potential with a negative pregnancy test (urine or serum)within 2 weeks prior to registration, preferably as close to the first dose as possible, and agrees to use adequate contraception.

Acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

An intrauterine device with a documented failure rate of less than 1% per year, Vasectomised partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female, Complete abstinence from sexual intercourse for 14 days before exposure to the investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product, Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).

* Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Exclusion Criteria:

* Known or suspected hypersensitivity reaction to the investigational compounds or incorporated substances.
* (Neo-)adjuvant therapy not containing a solvent based taxane.
* (Neo-)adjuvant therapy with nab-paclitaxel.
* Concurrent hormonal therapy for cancer.
* Life expectancy less than 3 months.
* Pre-existing peripheral neuropathy of > grade 2 (per CTCAE).
* Pre-existing grade 3 or 4 diarrhea.
* Presence of uncontrolled infection.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with the subject's safety, provision of informed consent, or compliance to study procedures.
* Concurrent specific systemic anti-tumor treatment or treatment with experimental compounds during study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 3 years

SECONDARY OUTCOMES:
Toxicity of the therapy | 3 years
  Number and percent of patients with Adverse Events (any Grade and Grade 3/4).
Clinical benefit rate (CBR) in patients with measurable disease | 3 years
Duration of response | 3 years
Progression-free survival (PFS) | 3 years
Overall survival (OS) | 3 years
SPARC expression rate of the tissue of the primary and/or metastatic tumor | 3 years
Compliance of the therapy | 3 years
  Number and percent of the patients with treatment modifications (dose delay / dose reduction / premature dicontinuation)

CONTACTS AND LOCATIONS:
Locations (1):
- GBG Forschungs GmbH, Neu-Isenburg, Germany